CLINICAL TRIAL: NCT05404464
Title: CITIC Xiangya Assisted Reproduction Data Repository: a Real Medical Environment Based Research Database
Brief Title: Construction of CITIC Xiangya Assisted Reproduction Data Repository
Acronym: CXARDR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Collaborators: Central South University (Other); West China Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LL-SC-2022-014
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Assisted Reproductive Technology; Infertility
Keywords: Population-based database; Registry; Infertile couple and offspring; Longitudinal study
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood, semen, follicular fluid and granulosa cell
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couples: Infertile couples who came to the hospital for ART treatment
  Interventions: Other: Different baseline characteristics and clinical management

INTERVENTIONS:
Other: Different baseline characteristics and clinical management — Personal history, basic diseases, stimulation plan, type of ART, transplantation strategy, etc.

SUMMARY:
Human Assisted Reproductive Technology (ART) has become a very effective and nearly irreplaceable clinical treatment for infertility, helping millions of women achieve fertility. However, ART may still have potential health risks to mothers and offspring. To better research and monitor the efficacy and safety of ART, the investigators established CXARDR based on the real medical data in Reproductive and Genetic Hospital of CITIC-Xiangya, which is the world's largest ART single treatment center. CXARDR covers the ART full-cycle treatment records since the hospital perfected its electronic medical record system in 2016, as well as biological samples from the CITIC-Xiangya Genetic Resource Bank. From the preoperative investigation of ART to the 1-year follow-up of ART offspring, CXARDR provides the details of the whole process of treatment and the follow-up outcomes of ART patients, making up for the gap in the data of reproductive and obstetric institutions. The huge biological samples with clinical information also provide more possibilities for in-depth basic researches in the field of reproduction and genetics.

During the past five years (January 2016 to November 2020), the CXARDR has accumulated data concerning more than 223,000 ART treatment cycles from 120,000 infertile couples. The CXARDR also links more than 180,000 blood samples, 65,000 follicular fluid samples, 80,000 semen samples, and 31,000 granulosa cell samples from 75,000 couples. The data volume is substantial with over 800 variables being documented, and most variables are designed as structured fields. The whole process of data access, data extraction, data processing and data analysis was conducted through a dedicated server inside the CITIC-Xiangya Data Center. All investigators cannot access sensitive information, are required to sign data confidentiality agreement, and need to be approved by the CITIC-Xiangya Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* All infertile couples undergoing ART treatment in our hospital (CITIC-Xiangya) were enrolled.

Exclusion Criteria:

* None.

Ages: 16 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile couples who received ART treatment in our hospital (CITIC-Xiangya).
Sampling Method: Probability Sample
Enrollment: 119590 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Cleavage rate | Up to 3 days after insemination
  The proportion of zygotes that cleave to become embryos on Day 2 (44 ± 1 h post-insemination) .
Implantation rate | Up to 30 days after transplantation
  The number of gestational sacs divided by the total number of embryos transferred, irrespective of whether a pregnancy was established.
Clinical pregnancy | Up to 30 days after transplantation
  A pregnancy diagnosed by ultrasonographic examination of at least one fetus with a discernible heartbeat.
Miscarriage | Up to 42 weeks after transplantation
  The spontaneous loss of an intrauterine pregnancy.
Live birth | Up to 42 weeks after transplantation
  The complete expulsion or extraction from a woman of a product of fertilization, after 20 completed weeks of gestational age.
Gestational age at birth | Up to 42 weeks after transplantation
  The age of a fetus is calculated by the best obstetric estimate determined by assessments which may include early ultrasound.
Birthweight | Up to 42 weeks after transplantation
  Birth weight should be collected within 24 hours of birth and assessed using a calibrated electronic scale with ten-gram resolution.
Height of offspring 1 year old | Up to 1 year after delivery
  Self-measurement
Weight of offspring 1 year old | Up to 1 year after delivery
  Self-measurement

SECONDARY OUTCOMES:
Embryo development rate | Up to 3 days after insemination
  The proportion of cleaved embryos at the 4-cell stage on Day 2 (44 ± 1 h post-insemination) or at the 8-cell stage on Day 3 (68 ± 1 h post-insemination) per normally fertilized oocyte.
1PN rate | Up to 2 days after insemination
  The proportion of inseminated oocytes with one pronucleus on Day 1 (17 ± 1 h post-insemination).
Blastocyst development rate | Up to 7 days after insemination
  The proportion of blastocysts observed at 116 ± 2 h post-insemination as a function of the number of normally fertilized oocytes.
Proportion of good blastocysts | Up to 7 days after insemination
  The proportion of blastocysts with a grade of "good" or higher.
Ectopic pregnancy | Up to 30 days after transplantation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization, or histopathology.
Gestational diabetes | Up to 30 weeks after transplantation
  By oral glucose tolerance test between 24 and 28 gestational weeks (fasting glucose ≥5.1 mmol/L, 1-h glucose ≥10.0 mmol/L, 2-h glucose ≥8.5 mmol/L; one abnormal result sufficient).
Gestational hypertension | Up to 42 weeks after transplantation
  Maternal systolic blood pressure ≥ 140 mmHg and (or) diastolic pressure ≥ 90 mmHg.
Major congenital anomaly | Up to 42 weeks after transplantation
  Structural, functional, and genetic anomalies, that occur during pregnancy, and identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or are life-threatening, or cause death.
Neonatal mortality | Up to 30 days after delivery
  Death of a live born baby within 28 days of birth.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ge, PhD, Study Director — Reproductive & Genetic Hospital of CITIC-XIANGYA Changsha, Hunan China

IPD SHARING:
Plan to Share IPD: Yes
According to the policy of CITIC-Xiangya Reproductive and Genetic Hospital,research institutions could apply for data access by submitting a formal study protocol, subjected to approval by the hospital academic committee. Ethical review and research registration are mandatory for all studies.